CLINICAL TRIAL: NCT03545672
Title: EARLY Identification of MYOcardial Impairment in Primary Biliary Cholangitis
Brief Title: Early Identification of Myocardial Impairment in PBC
Acronym: EARLY-MYO-PBC
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201709P
Record Dates: First submitted 2018-02-01; First posted 2018-06-04 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-03

CONDITIONS: Primary Biliary Cholangitis; Cardiovascular Abnormalities
Keywords: Primary Biliary Cholangitis; Cardiac impairment; Cardiovascular Magnetic Resonance
MeSH Terms: conditions — Liver Cirrhosis, Biliary; Cardiovascular Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PBC group: Patients have a definite PBC diagnosis.
  Interventions: Diagnostic Test: CMR examination
- Control group: The healthy volunteers.
  Interventions: Diagnostic Test: CMR examination

INTERVENTIONS:
Diagnostic Test: CMR examination — After recruiting participants and collecting the baseline information, a CMR scan and a post-processed imaging procedure will be carried on in order to detect the cardiac impairment.

SUMMARY:
Primary biliary cholangitis (PBC) is a chronic inflammatory liver disease leading to cirrhosis. Researches reported patients with PBC may involve abnormalities on skeleton, thyroid and exocrine glands. However, whether this autoimmune disease would cause cardiac impairment is scarcely investigated. Cardiovascular Magnetic Resonance(CMR) is recently developed as a reliable modality to evaluate the cardiac tissue characteristics and functions. This study aims to investigate the cardiac status in PBC patients based on CMR.

DETAILED DESCRIPTION:
Primary biliary cholangitis (PBC) is a progressive and uncommon inflammatory autoimmune cholesteric liver disease，which will contribute to cirrhosis. Symptoms and course of primary biliary cholangitis can be diverse, wherefore the targets of the current treatment are focused on the prevention of end-stage liver disease. Researches reported patients with PBC may involve abnormalities on skeleton, thyroid and exocrine glands. However, whether this autoimmune disease would cause cardiac impairment is scarcely investigated. From our clinical practice, the cardiac structural abnormal can be found in certain patients with PBC detected by cardiovascular magnet resonance (CMR). CMR is the primary and emerging imaging modality for myocardial tissue characterization, and it is recommended as a gold standard for functional imaging and assessment. This three-center, multi-modality, prospective observational study plans to identify the type and the severity of cardiac changes in PBC.

ELIGIBILITY:
Inclusion Criteria for PBC group:

* Age between 18-80 years old.
* Definite primary biliary cirrhosis diagnosis which is consistent with European Association for the Study of the Liver (EASL) [Clinical Practice Guidelines: The diagnosis and management of patients with primary biliary cholangitis (2017)]. The following three diagnostic factors, at least meet two:

  1. History of elevated alkaline phosphatase (ALP) levels;
  2. Liver biopsy consistent with PBC;
  3. Positive antimitochondrial antibodies (AMA) or specific antinuclear antibodies;
* Providing written informed consent

Exclusion Criteria:

* History or presence of other concomitant liver disease including:

  1. cirrhosis or viral hepatitis;
  2. Inherited metabolic liver disease;
  3. Drug-induced liver injury;
  4. Other systemic disease inducing liver change.
* Subjects with life expectancy < 6 months.
* Subjects with known ischemic/non-ischemic cardiomyopathy or abnormal in cardiac-related examinations.
* Subjects with standard metallic contraindications to CMR (i.e., estimated glomerular filtration rate < 30 ml/min/1.73 m2, New York Heart Association functional capacity class IV)

Inclusion Criteria for Control group:

* Absence of known systemic diseases
* Normal examinations in CMR/Echo/ECG
* Age between 18-80 years old.
* Providing written informed consent

Exclusion Criteria:

* Subjects with known heart disease including:

  1. Documented coronary artery disease;
  2. Ischemia/non-ischemia cardiomyopathy;
  3. Other systemic disease inducing heart change.
* Subjects with known liver disease including:

  1. Viral hepatitis;
  2. Inherited metabolic liver disease;
  3. Drug-induced liver injury;
  4. Other systemic disease inducing liver change.
* Subjects with standard metallic contraindications to CMR

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive subjects from three centers were prospectively enrolled into 2 cohorts between September 2017 and April 2019. The cohorts were divided as follows: the PBC patients group and the control group.
Sampling Method: Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meng Jiang, MD, Study Chair — RenJi Hospital, School of Medicine, Shanghai Jiantong University; Xiong Ma, MD,PhD, Study Chair — RenJi Hospital, School of Medicine, Shanghai Jiantong University
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jiang P, Feng Z, Sheng L, Hu C, Ma X, Zhang S, Wu L, Xiao X, Wang Q, Guo C, Qiu D, Fang J, Xu J, Gershwin ME, Jiang M, Ma X, Pu J. Morphological, Functional, and Tissue Characterization of Silent Myocardial Involvement in Patients With Primary Biliary Cholangitis. Clin Gastroenterol Hepatol. 2022 May;20(5):1112-1121.e4. doi: 10.1016/j.cgh.2021.08.035. Epub 2021 Aug 28. PMID 34461299

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a prospective, three-center, cardiac imaging observational study. The study was open for recruitment between September 2017 and January 2019. The first participant was enrolled on October 23, 2017 and last participant was enrolled on January 8, 2019
Pre-assignment Details: Of 119 enrolled participants. 112 participants were included and randomized to observational study group.
Groups:
- PBC Group: Patients have a definite PBC diagnosis.
  Cardiac Magnetic Resonance (CMR) examination: After recruiting participants and collecting the baseline information, a CMR scan and a post-processed imaging procedure will be carried on in order to detect the cardiac impairment.
Period: Overall Study
Arm/Group | PBC Group | Control Group
Started | 60 | 59
Completed | 56 | 56
Not Completed | 4 | 3
Not completed — Uncertain diagnosis | 2 | 1
Not completed — Protocol Violation | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PBC Group | Control Group | Total
Number analyzed (Participants) | 56 | 56 | 112
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 52 [47 to 56] | 48 [29 to 57] | 52 [38 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 46 | 96
  Male | 6 | 10 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 56 | 56 | 112
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 23 [20 to 25] | 23 [20 to 26] | 23 [20 to 25]
Heart rate [Median (Inter-Quartile Range); unit: beats/min] | 71 [70 to 80] | 71 [64 to 80] | 71 [67 to 80]
NYHA classification of heart failure class III-IV [Count of Participants; unit: Participants] — "The New York Heart Association (NYHA) Classification of Heart Failure is used to classify the severity of heart failure or heart function based on daily activities. In this study, it was defined as follows: Class I-II: No or only slight limitation of physical activity. Ordinary activity does not cause undue fatigue, palpitation, or dyspnea.
  Class III-IV: Marked limitation of physical activity, or inability to carry on any activity without discomfort."
  Participants | 0 | 0 | 0
Other autoimmune diseases [Count of Participants; unit: Participants] | 5 | 0 | 5
Hemoglobin [Median (Inter-Quartile Range); unit: g/L] | 124 [111 to 132] | 133 [124 to 142] | 129 [119 to 137]
Platelet [Median (Inter-Quartile Range); unit: platelets *10^9/L] | 173 [98 to 253] | 225 [202 to 251] | 200 [154 to 251]
Serum creatinine [Median (Inter-Quartile Range); unit: μmol/L] | 55.1 [49 to 63.8] | 60.5 [52 to 70.8] | 58 [50 to 68]
Native myocardium T1 mapping [Median (Inter-Quartile Range); unit: msec] — T1 mapping is a magnetic resonance imaging (MRI) technique used to measure the longitudinal relaxation time (T1) of tissues in the heart. It can provide quantitative information about the myocardial tissue composition, such as fibrosis (scarring of the heart tissue), edema (swelling due to fluid retention), and amyloidosis (deposition of amyloid proteins).
  msec | 1317 [1285 to 1356] | 1284 [1268 to 1317] | 1299 [1274 to 1329]
T2 mapping [Median (Inter-Quartile Range); unit: msec] | 50 [47 to 53] | 48 [46 to 50] | 48 [46 to 51]
Volume parameters [Median (Inter-Quartile Range); unit: mL] — LVEDV: Left ventricular end-diastolic volume; LVESV: Left ventricular end-systolic volume
  mL
    LVEDV | 103 [94 to 120] | 107 [95 to 118] | 105 [94 to 119]
    LVESV | 27 [21 to 31] | 31 [24 to 37] | 28 [23 to 35]
Left Ventricular Ejection Fraction [Median (Inter-Quartile Range); unit: %] | 75 [71 to 79] | 69 [67 to 72] | 72 [69 to 77]
Myocardium Strain [Median (Inter-Quartile Range); unit: %] — Myocardial strain refers to the deformation (stretching, thickening, or shortening) of heart muscle (myocardium) during the cardiac cycle, compared to its original shape. Global longitudinal strain (GLS) measures the percentage change in the length of the myocardial fibers (heart muscle cells) during the cardiac cycle. Global Circumferential Strain (GCS) measures the degree of myocardial deformation in the circumferential direction around the short axis of the heart.
  %
    GLS | -18.4 [-20 to -16.7] | -17.4 [-18.8 to -15.3] | -17.8 [-19.3 to -15.9]
    GCS | -22.5 [-24 to -21.4] | -20.8 [-22.6 to -19.2] | -21.8 [-23.4 to -19.8]
T2-STIR positive [Count of Participants; unit: Participants] — T2-STIR (Short Tau Inversion Recovery) positive indicate the myocardium edema.
  Participants | 12 | 1 | 13
LGE positive [Count of Participants; unit: Participants] — Late Gadolinium Enhancement (LGE) is used to detect and visualize myocardial scarring or fibrosis.
  Participants | 20 | 5 | 25

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Cardiac Events
Description: All PBC patients are followed up through telephone or by retrieving outpatient medical record systems. Cardiac events include: 1. cardiac death; 2. myocardial infarction; 3. hospitalization for unstable angina.
Time Frame: 7 months after first CMR scanning
Measure: Count of Participants; unit: Participants
Arm/Group | PBC Group | Control Group
Number analyzed (Participants) | 56 | 56
Participants
  Cardiac death | 0 | 0
  Myocardial infarction | 0 | 0
  Hospitalization for unstable angina | 0 | 0
Statistical Analysis 1: Comparison: PBC Group vs Control Group; Test type: Superiority; p = 0.001, Chi-squared — The threshold for statistical significance was p=0.05

2. Primary Outcome: Quantitative Assessment in Cardiac Injury
Description: T1 mapping-derived extracellular volumes (ECV) were used to detect changes in the myocardium interstitial matrix. ECV was calculated according to the ECV formula consist of T1 mapping value.
Time Frame: within 2 days of CMR scan
Measure: Median (Inter-Quartile Range); unit: percentage of interstitial matrix
Arm/Group | PBC Group | Control Group
Number analyzed (Participants) | 56 | 56
percentage of interstitial matrix | 30 [27 to 32] | 26 [25 to 27]
Statistical Analysis 1: Comparison: PBC Group vs Control Group; Test type: Superiority; p < 0.01, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse Event data were collected after first completion of cardiac magnetic resonance in 1 year.
Arm/Group | PBC Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/56
Other Adverse Events (participants affected / at risk) | 0/56 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-25): https://cdn.clinicaltrials.gov/large-docs/72/NCT03545672/Prot_SAP_000.pdf